CLINICAL TRIAL: NCT04054232
Title: A Randomized Controlled Trial to Evaluate an EHR-based PAD Screening Tool
Brief Title: Evaluation of an Electronic Health Record-based Screening Tool for Peripheral Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elsie Ross, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 52645; 1K01HL148639 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients with a high risk of having undiagnosed PAD will be identified using an EHR-based PAD screening tool. Fifty total patients meeting inclusion criteria will be randomized to either the intervention arm - primary treating physician notified about high risk of undiagnosed PAD - or the control arm - no notification provided. Physician notification will include suggestions to refer the patient to vascular medicine and/or order ankle brachial index (ABI) testing. If a patient is found to have PAD diagnosed by ABI the patient and provider will be notified and provided guidelines from the American Heart Association regarding management of PAD.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator will not be involved in the randomization process or in the process of collecting outcome data. Once data collection is complete, an independent investigator not involved in the trial will confirm study endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR Alert (Experimental): Twenty-five participants who are flagged by the screening tool as having high risk of undiagnosed peripheral artery disease (PAD) will be randomized to have their primary care physician receive an electronic health record message regarding their high risk of having PAD and a recommendation will be made to have the participant referred for non-invasive testing called Ankle Brachial Index (ABI) testing to confirm diagnosis. For individuals who undergo ABI testing and are confirmed to have PAD, they and their physicians will be provided with American Heart Association Guidelines for the management of PAD. Each participant's medical record will be reviewed for 6 months to evaluate for referral for ABI testing, referral to cardiovascular specialists (vascular medicine, vascular surgery or a cardiologist), and for initiation of new cardiovascular related medications such as an antiplatelet, statins, or anti-hypertensive medications.
  Interventions: Other: High PAD risk Alert
- No EHR Alert (No Intervention): Twenty-five participants who are flagged by the screening tool as having high risk of undiagnosed peripheral artery disease (PAD) will be randomized to the control arm and they nor their physicians will be alerted of their status for 6 months. Each participant's medical record will be reviewed for 6 months to evaluate for referral for ABI testing, referral to cardiovascular specialists (vascular medicine, vascular surgery or a cardiologist), and for initiation of new cardiovascular related medications such as an antiplatelet, statins, or anti-hypertensive medications. At the end of 6 months of observation, the primary care physician's of control participants will receive the same alert as participants in the intervention arm.

INTERVENTIONS:
Other: High PAD risk Alert — In this message sent via the electronic health record, a participant's primary care physician will receive a message that details the following:
  1. Participant flagged as having a high risk of peripheral artery disease based on their electronic health record data
  2. What peripheral artery disease is and why diagnosis may be important
  3. Recommendation to refer to a vascular medicine specialist or order ankle brachial index for definitive diagnosis
  4. The option to opt out if the potential participant is not deemed a candidate for inclusion in the study with a short explanation of why the potential participant should not be included.
  Arms: EHR Alert

SUMMARY:
This protocol represents a pilot randomized-controlled trial evaluating the effect of an electronic health record (EHR)-based peripheral artery disease (PAD) screening tool on rates of new non-invasive testing, diagnosis and treatment of PAD over a 6-month period. An EHR-based PAD screening tool will be applied to the Stanford EHR, which will generate a group of patients of varying risks of having undiagnosed PAD. Patients with the highest risk of having undiagnosed PAD will then be evaluated for inclusion in this study. 1:1 randomization will be performed on a consecutive basis until study enrollment is completed (25 patients per arm).

Physicians of patients randomized to the intervention arm will be sent notification via an EHR message detailing the patient's risk of undiagnosed PAD and suggestions for referral to vascular medicine for risk assessment and/or non-invasive ankle brachial index (ABI) testing. The primary outcome is number of patients receiving ABI testing for PAD at 6 months, with secondary outcomes including number of new PAD diagnoses, number of new referrals to cardiovascular specialists (vascular medicine, vascular surgery, and/or cardiology) and number of patients receiving initiation of new cardiovascular medications (anti-platelet agents, statins, and/or antihypertensive agents).

ELIGIBILITY:
Inclusion Criteria:

* Are 50-85 years old
* Currently an outpatient, actively obtaining care at Stanford
* Have at least 1 year of data within the Stanford EHR (including at least 2 clinical visits)
* Have no prior diagnosis of peripheral artery disease as determined by no chart term mentions or ICD-9/10 codes in their EHR data

Exclusion Criteria:

* Have less than 1 year of data available or less than 2 clinical visits at Stanford
* Enrolled in a previous related study
* Receiving treatment for a potentially terminal condition
* Prior diagnosis of peripheral artery disease by ICD code or term mention in their EHR data.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
New referral for ankle brachial index testing | 6 months after randomization
  Number of new orders/referrals to obtain non-invasive diagnosis of peripheral artery disease with ankle-brachial index in each arm 6 months after randomization.

SECONDARY OUTCOMES:
New PAD diagnosis | 6 months after randomization
  Number of patients newly diagnosed with peripheral artery disease in each arm 6 months after randomization.
New referral to cardiovascular specialist | 6 months after randomization
  Number of new referrals to cardiovascular specialists (vascular medicine, vascular surgery and/or cardiology) in each arm 6 months after randomization.
New prescriptions for guideline-recommended medications | 6 months after randomization
  Number of new prescriptions given for antiplatelet agent, statin, and/or antihypertensive agents in each arm 6 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Ross, MD, MSc, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.